CLINICAL TRIAL: NCT03420287
Title: Evaluation of Mineralized Plasmatic Matrix Prepared From Allogenic Bone Graft in Alveolar Cleft Closure: A Prospective Randomized, Triple Blinded, Parallel Clinical Trial
Brief Title: Evaluation of MPM Prepared From Allogenic Bone Graft in Alveolar Cleft Closure: A Prospective Randomized Clinical Trial
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Salah, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-01-02
Record Dates: First submitted 2018-01-28; First posted 2018-02-05 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-01

CONDITIONS: Cleft; Alveolar Process

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MPM prepared from allogenic bone graft (Experimental): All patients in this group will receive MPM prepared from allogenic bone graft
  Interventions: Combination Product: MPM Prepared From Allogenic Bone Graft
- Autogenous bone graft group (Active Comparator): All patients in this group will receive autogenous bone graft only
  Interventions: Other: Autogenous bone

INTERVENTIONS:
Combination Product: MPM Prepared From Allogenic Bone Graft — patients will receive a sticky bone which prepared by mixing the the growth factors of the patient with allogenic bone graft for cleft closure
  Arms: MPM prepared from allogenic bone graft
Other: Autogenous bone — patients will receive an autogenous bone graft from anterior iliac crest for cleft closure
  Arms: Autogenous bone graft group

SUMMARY:
The aim of this trial is to figure out the efficiency of Mineralized Plasmatic Matrix prepared from allogenic bone graft on cleft alveolus and oro-nasal fistula closure, adequate bone volume and acceptable density at the site of grafting.MPM might improve the physiological properties of allogenic bone graft and facilitate its handling and application during surgical grafting.This might decrease the need of the second surgical site for harvesting autogenous bone to be grafted with its all complications and hurdles.This trial will help the practitioners in taking the decision of using the MPM prepared from allogenic bone in alveolar cleft closure or not.

DETAILED DESCRIPTION:
Alveolar bone grafting will be performed at 6 to 12 years of age as following :

Group (A):Will undergo grafting with anterior iliac crest bone,(Control group). Group (B):Will undergo grafting with Mineralized Plasmatic Matrix prepared from allogenic bone graft (study group).

In all patients, this will be the first bone graft to be placed in the alveolar cleft. All patients will be monitored clinically and radiographically (by cone beam C.T) for up to 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral alveolar cleft patients

Exclusion Criteria:

* patients with previous failed alveolar cleft grafting procedure.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Oro-nasal Fistula | 6 months
  it will be assessed visually and by questionnaire with binary measuring unit (present or not).• Examination of oro-nasal Fistula will be done by using the following diagnostic criteria: 1.Air escape from the opening when patient blows his/her nose.
  2.An obvious communication between the opening and floor of the nasal cavity. 3.Unobstructed penetration of Guttapercha through the opening into the nasal cavity.
  4.Hypernasality of voice due to audible nasal air escape during speech. 5.Nasal regurgitation of fluids. 6.Food lodgement into nasal cavity with risk of rhinitis .

SECONDARY OUTCOMES:
C.T analysis of secondary bone grafts | 6 months
  it will be assessed by Chelsea Scale which radio-graphically analyzing the position of the bone tissue in relation to the teeth adjacent to the cleft and separating the images into 6 categories: A,B,C,D, E,F.
  Bone grafts of types A,B and C according to the Chelsea scale were considered satisfactory, whereas the other types were considered unsatisfactory
Donor site long standing pain | 6 months
  it will be assessed by Numeric Rating Scale (NRS).Numeric Rating ScaleUsing the NPRS which is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The common format is a horizontal bar or line.
  (NRS).0 means no pain, 5 means moderate pain and 10 means worst possible pain.